CLINICAL TRIAL: NCT06714578
Title: Construction of a Risk Screening Tool for New Psychoactive Substance Misuse Among Adolescents and Young Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, Principal Investigator, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: L2024SYSU-HL-039
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Drug Misuse; Addiction
MeSH Terms: conditions — Drug Misuse; Behavior, Addictive | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire and Physical Exam — The investigators use questionnaire to assess biological factors (sleep quality, externalizing problem behavior, prosocial tendencies, sensation seeking, and hedonic hunger), psychological factors (risk awareness of drug misusing, indulgence of drug misusing, self-efficacy of drug misusing, and ACEs), and social factors (whether work in a special place, whether have drug-addicts around, cognition of traditional drug types, and cognition of NPS types) and demographic data

SUMMARY:
The goal of this observational study is to construct a risk tool available for screening young adults and adolescents at high risk of drug misuse and provides a chance for early intervention to young adults and adolescents at high risk of drug misuse, which prevent the onset and development of drug addiction in the future.The main question it aims to answer is:

1. Explore the occurrence and influencing factors of new psychoactive substance misuse among young adults and adolescents;
2. Construct a risk prediction model for new psychoactive substance misuse among young adults and adolescents and conduct internal verification of the model;
3. Based on the results of the prediction model, select the optimal model to initially form a concise scale "Screening Tool for the Risk of New Psychoactive Substance Misuse among Young Adults and Adolescents";
4. Conduct external verification of the tool, and revise and improve the screening tool, form the final version of the screening tool, and verify the application performance of the screening tool.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults who were aged 14-35 years;
* Adolescents and young adults could read and communicate in Chinese were invited to participate in this study

Exclusion Criteria:

* Adolescents and young adults who were unable to complete the questionnaire due to physical or psychological reasons.

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents and young adults aging 14-35 years old
Sampling Method: Non-Probability Sample
Enrollment: 1035 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Perceived risks associated with drug abuse | baseline
  Perceived risks associated with drug abuse developed by the Hong Kong Security Bureau's Narcotics Division is adopted (https://www.nd.gov.hk/tc/beat_questions_2010R2.html). The scale consists of 12 questions and uses a 5-point Likert scale (1 = Strongly Disagree, 2 = Disagree, 3 = Unsure, 4 = Agree, 5 = Strongly Agree). The total score ranges from 12 to 60, with a higher score indicating a greater awareness of drug use risks. In this study, the Cronbach's α coefficient for the Chinese version of this scale is 0.931.
Pittsburgh Sleep Quality Index (PSQI) | baseline
  The Pittsburgh Sleep Quality Index was developed by Buysse et al. [14], and the Chinese version was translated and revised by Xianchen Liu et al. in 1996 [15]. It has been confirmed that the PSQI is suitable for evaluating sleep quality in patients with mental disorders and the general population in China. This scale consists of 19 self-reported items and 5 observer-rated items, of which the 19th self-reported item and the 5 observer-rated items are not included in the scoring. The 18 items comprise seven factors: sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. Each component is scored on a scale from 0 to 3, with a total score range from 0 to 21. A higher score indicates poorer sleep quality. In this study, the overall Cronbach's α coefficient for the Chinese version of the scale across the seven factors was 0.716.
Prosocial Tendencies Measure (PTM) | baseline
  The Chinese version of the Prosocial Tendencies Measure was revised by Yu Kou, Huifang Hong et al. in 2007 [16]. This scale consists of 26 items, encompassing six dimensions: public, anonymous, altruistic, compliant, emotional, and urgent. It uses a 5-point Likert scale for scoring (1 = very unlike me, 2 = somewhat unlike me, 3 = neutral, 4 = somewhat like me, 5 = very like me). The total score ranges from 26 to 130, with higher scores indicating greater prosocial tendencies. In this study, the Cronbach's α coefficient for the Chinese version of the scale was 0.957, with the Cronbach's α coefficients for the six dimensions of public, anonymous, altruistic, compliant, emotional, and urgent being 0.824, 0.877, 0.845, 0.849, 0.855, and 0.791, respectively.
Achenbach Youth Self Report (YSR) | baseline
  The Youth Self Report (YSR), developed by Achenbach et al. [17], was used in its 2001 version. The Chinese version was translated and revised by Wang Runcheng et al.[18] in 2013. The questionnaire is divided into 8 factors (Anxiety/Depression, Withdrawn/Depressed, Somatic Complaints, Social Problems, Thought Problems, Attention Problems, Delinquent Behavior, Aggressive Behavior) and an "Other Problems" item. The Delinquent Behavior and Aggressive Behavior factors together constitute the externalizing symptom group and are widely used to measure externalizing problem behaviors in adolescents. The Delinquent Behavior factor includes 15 items, and the Aggressive Behavior factor includes 17 items, using a three-point scoring scale (0 = not at all true, 1 = somewhat true, 2 = very true). The total score for the two factors ranges from 0 to 96, with higher scores indicating more severe externalizing problem behaviors. In this study, the Cronbach's α coefficients for the Delinquent Behavior
Brief Sensation Seeking Scale for Chinese (BSSS-C) | baseline
  The 8-item Brief Sensation Seeking Scale developed by Hoyle et al.[19] was utilized, with the Chinese version translated and revised by Xinguang Chen et al.[20] in 2013 to measure personality traits related to sensation seeking. This scale comprises 8 items, encompassing four dimensions: Lack of Self-Control, Pursuit of Novelty, Difficulty Tolerating Monotony, and Pursuit of New Experiences. A five-point Likert scale was used for scoring (1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree). The total score ranges from 8 to 40, with higher scores indicating higher levels of sensation seeking. In this study, the Cronbach's α coefficient for the Chinese version of the scale was 0.855.
Power of Food Scale (PFS) | baseline
  The Power of Food Scale developed by Lowe et al.[21] was employed, with the Chinese version translated and revised by Han Xiao, Jianwen Song, Xinni Han et al.[22] in 2023, to measure the level of hedonic hunger. The scale consists of 15 items, which include three dimensions: Food Availability, Food Presence, and Food Taste, utilizing a five-point Likert scale for scoring (1 = I disagree, 2 = I somewhat agree, 3 = I somewhat agree, 4 = I fairly agree, 5 = I completely agree). The total score ranges from 15 to 75, with higher total scores indicating a greater level of hedonic hunger. In this study, the Cronbach's α coefficient for the Chinese version of the scale was 0.940, and the Cronbach's α coefficients for the three dimensions (Food Availability, Food Presence, Food Taste) were 0.866, 0.858, and 0.863, respectively.
Permissive attitude towards drug abuse | baseline
  Permissive attitude towards drug abuse developed by the Hong Kong Security Bureau's Narcotics Division is adopted (https://www.nd.gov.hk/tc/beat_questions_2010R2.html). The scale consists of 21 questions and uses a 5-point Likert scale (1 = Strongly Disagree, 2 = Disagree, 3 = Unsure, 4 = Agree, 5 = Strongly Agree). The total score ranges from 21 to 105, with a higher score indicating a higher tolerance attitude towards drug use. In this study, the Cronbach's α coefficient for the Chinese version of this scale is 0.966.
Refusal Self-Efficacy Scale (Self-Efficacy List for Drug Users, SELD) | baseline
  The Refusal Self-Efficacy Scale developed by Gerdien et al.[23] is adopted (Self-Efficacy List for Drug Users, SELD), with the Chinese version translated and revised by Liuna Geng et al.[24], used to measure refusal self-efficacy regarding drugs. The scale consists of 17 questions encompassing three dimensions: environmental factors, negative emotions, and positive emotions, using a 5-point Likert scale (1 = Very Easy to Refuse, 2 = Easy to Refuse, 3 = Unsure, 4 = Somewhat Difficult to Refuse, 5 = Very Difficult to Refuse). The total score ranges from 17 to 85, with a higher score indicating lower refusal self-efficacy. In this study, the Cronbach's α coefficient for the Chinese version of this scale is 0.961, and the Cronbach's α coefficients for the three dimensions (environmental factors, negative emotions, positive emotions) are 0.901, 0.928, and 0.937, respectively.
Adverse childhood experiences, ACEs | baseline
  The Adverse Childhood Experiences Scale developed by the Kaiser-CDC laboratory is adopted to investigate various adverse events experienced by subjects before the age of 18[25]. The scale includes three dimensions: abuse, neglect, and family dysfunction, with a total of 10 items. Each item offers two response options: "Yes" and "No." A "Yes" response is scored as 1 point, while a "No" response is scored as 0 points. The total score is the sum of the scores from each item, reflecting the number of adverse childhood experiences. The total score ranges from 0 to 10, with a higher score indicating more adverse childhood experiences. In this study, the Cronbach's α coefficient for the Chinese version of this scale is 0.760.
Peers drug-misuse situation | baseline
  It is a binary outcome. The investigators will ask for question that "Are there peers around you engage in drug use?" And the participants are supposed to answer "yes" or "no"
Work experiences in special venues | baseline
  The investigators will ask for question that "Do you have any work experience in special venues such as bars or nightclubs?" And the participants are supposed to choose the special venues they used to work including "Bar", "Internet cafe", "Ballroom", "Nightclub", "KTV", "Disco", "Leisure clubhouse", "Agriturismo" or choose "None of the above" if they have never work in such special venues.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China